CLINICAL TRIAL: NCT07024758
Title: Comparative Effectiveness of Internet-based Versus Parent-Coached Cognitive-Behavioral Therapy For Children and Adolescents With Anxiety and OCD
Acronym: ASTRO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Eric A Storch, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-57367
Record Dates: First submitted 2025-06-03; First posted 2025-06-17 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Obsessive Compulsive Disorder (OCD); Anxiety Disorder of Childhood or Adolescence; Social Anxiety Disorder of Childhood; Generalized Anxiety Disorder (GAD); Separation Anxiety Disorder; Panic Disorder; Panic Attacks; Panic Disorder (With or Without Agoraphobia); Phobia, Specific
Keywords: Obsessive-compulsive disorder; anxiety; cognitive-behavioral therapy; children; adolescents
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Generalized Anxiety Disorder; Anxiety, Separation; Panic Disorder; Phobia, Specific; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Children (N=174) ages 7-17 will be randomized into one of two conditions.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor is blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parent Coached Exposure Therapy (PCET) (Active Comparator): Parent Coached Exposure Therapy (PCET) consists of 12 weekly individual sessions that are attended by the therapist, child, and parent. Sessions will follow the cognitive behavioral therapy model of childhood anxiety disorders, wherein safety behaviors and avoidance reinforce anxiety, explains the rationale of exposure, and begins developing an exposure hierarchy with the family. Sessions will include psychoeducation, developing an exposure hierarchy, carrying out in-session exposures, and assigning exposures in between sessions.
  Interventions: Behavioral: Parent Coached Exposure Therapy
- Family-Based Internet-Based CBT Group (iCBT) (Active Comparator): One half of participants will be randomized to receive iCBT. Each week of treatment, the parent will be encouraged to read the corresponding materials on the Baylor College of Medicine (BCM) webpage, complete accompanying worksheets, and guide their child through completing activities in the child-facing materials, with support from a therapist (7 45-minute supportive therapy sessions). One core aspect of treatment will be parents leading their child through graduated exposure. Exposures, a hallmark of CBT for anxiety, are used to gradually and repeatedly confront feared stimuli. For example, exposure therapy for a child fearful of dogs may begin with looking at pictures of dogs and standing across the park from a dog on a leash, to eventually petting a dog. All relevant information regarding parent-led exposures will be detailed in the treatment materials, and therapists will review with parents via email and/or video-conferencing sessions.
  Interventions: Behavioral: Family Based, Internet-Based Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Parent Coached Exposure Therapy — Parent-based cognitive behavioral therapy with guidance from a therapist
  Arms: Parent Coached Exposure Therapy (PCET)
Behavioral: Family Based, Internet-Based Cognitive Behavioral Therapy — Family-based cognitive behavioral therapy employing internet-delivered modules and videos
  Arms: Family-Based Internet-Based CBT Group (iCBT)

SUMMARY:
Anxiety disorders in children and adolescents are common and confer significant disability. Cognitive behavioral therapy (CBT) is the recommended treatment for youth with anxiety, yet many families cannot access CBT due to cost, practicalities of attending in-person treatment sessions, and a shortage of trained providers, especially in rural areas. To combat these barriers, other treatment methods have been developed.

Previous research has shown that family-based, internet-delivered CBT (iCBT) for anxiety and OCD in youth has shown a significant reduction in anxiety symptoms. Parent-coached exposure therapy (PCET) focuses entirely on teaching parents and youth together how to address anxiety through the completion of in-session parent-coached exposures and assigning parent-coached exposure as homework in between sessions.

Although both iCBT and PCET show positive results in treating pediatric anxiety in comparison to standard-care CBT, little is known about the comparative efficacy of iCBT and PCET.

This research is being done to understand the comparative effectiveness of two different types of cognitive-behavioral therapy (CBT) for treating anxiety or OCD in youth.

DETAILED DESCRIPTION:
Anxiety disorders in children and adolescents are common and confer significant disability. Without treatment, anxiety remains chronic and contributes to increased risk for later suicidality, mood, and substance use disorders. Cognitive behavioral therapy (CBT) is the recommended treatment for youth with anxiety, yet many families cannot access CBT due to cost, practicalities of attending in-person treatment sessions, and a shortage of trained providers, especially in rural areas. To combat these barriers, other treatment methods have been developed.

Low intensity telehealth delivery of services is a promising method to improve access to care for youth with anxiety and their families, given its reachability to a wider range of areas (e.g., rural/underserved) and its ability to minimize practical barriers (e.g., treatment could be delivered to the youth's home without need for travel), and reduce stigma (e.g., parents do not need to visit mental health clinics). Previous research has shown that family-based, internet-delivered CBT (iCBT) for anxiety and OCD in youth has shown a significant reduction in anxiety symptoms.

Parent-coached exposure therapy (PCET) focuses entirely on teaching parents and youth together how to address anxiety through the completion of in-session parent-coached exposures and assigning parent-coached exposure as homework in between sessions. PCET is designed to treat anxiety more effectively and efficiently, allowing for fewer sessions and greater symptom remission than standard-care CBT.

Although both iCBT and PCET show positive results in treating pediatric anxiety in comparison to standard-care CBT, little is known about the comparative efficacy of iCBT and PCET.

This research is being done to understand the comparative effectiveness of two different types of cognitive-behavioral therapy (CBT) for treating anxiety or OCD in youth.

ELIGIBILITY:
Inclusion Criteria:

* The child is between the ages of 7 to 17 years inclusive at enrollment.
* The child has clinically significant symptoms of anxiety and/or OCD, as indicated by a score of 12 or higher on the Pediatric Anxiety Rating Scale (PARS).
* The child is appropriate for anxiety-focused treatment (e.g., anxiety or OCD is the primary or co-primary problem as diagnosed using the DIAMOND-KID).
* One parent/guardian is able and willing to participate in assessment and treatment (e.g., has sufficient English fluency, the decisional capacity to participate, and can commit to treatment duration).
* The participating parent/guardian lives with their child at least 50% of the time per self-report.
* Both parent and child can read and understand English.
* The participant has an IQ above 69, based on the KBIT-2, another valid test or clinician judgement (e.g., a previous assessment conducted, and report shared with study team).
* Participants must be in the state of Texas for treatment sessions/assessments.

Exclusion Criteria:

* The child has a diagnosis of a lifetime psychotic disorder and/or conduct disorder.
* The child has significant, current and active suicidality/homicidality and/or self-injury requiring medical intervention.
* The child has limited verbal communication abilities (e.g., no independent verbal communication).
* The child is receiving concurrent psychotherapy with anxiety and/or OCD as the primary focus. They can pause ongoing therapy to enroll.
* The child has initiated new antidepressant medication within 12-weeks of assessment (4-weeks for stimulants/benzodiazepines/antipsychotics) or during therapy.
* The child has changed psychotropic medication dosage within 4-weeks of assessment (2-weeks for stimulants/benzodiazepines/antipsychotics) or during therapy.
* The child requires a higher level of care than can be provided through the study (e.g., significant, current suicidal ideation).

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 174 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in clinician-rated child anxiety severity (PARS) throughout the past week. | baseline (before treatment or week 1), post-treatment (week 14), 1 month follow up (Week 18)
  Each item is scored on a 0 to 5 scale (higher scores correspond to greater severity), yielding a total between 0 and 30.

SECONDARY OUTCOMES:
Diagnostic Interview for Anxiety, Mood, and OCD and Related Neuropsychiatric Disorders (DIAMOND) with Clinical Severity Ratings | baseline (before treatment or week 1), post-treatment (week 14), 1 month follow up (Week 18)
  Clinician-rated diagnostic interview that includes current anxiety disorders, mood disorders, obsessive-compulsive disorder, and related neuropsychiatric disorders. Each diagnostic category is coded as present or absent based on symptom criteria and severity scale. Severity scales are scored on a 1-7 scale (1 = normal; 7 = extreme) and are based on current level of distress and impairment (within the past month).
Clinical Global Impression-Severity | baseline (before treatment or Week 1), during treatment (on average 14 weeks), post-treatment (Week 14), 1 month follow up (Week 18)
  Clinician-rated child psychopathology severity rating. A single item is scored 0-6 (0= no illness; 6= extremely severe symptoms).

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Whiteside SPH, Biggs BK, Geske JR, Gloe LM, Reneson-Feeder ST, Cunningham M, Dammann JE, Brennan E, Ong ML, Olsen MW, Hofschulte DR. Parent-coached exposure therapy versus cognitive behavior therapy for childhood anxiety disorders. J Anxiety Disord. 2024 Jun;104:102877. doi: 10.1016/j.janxdis.2024.102877. Epub 2024 May 18. PMID 38788593
- [Background] Guzick AG, Schneider SC, Perozo Garcia AB, Kook M, Greenberg RL, Riddle D, McNeel M, Rodriguez-Barajas S, Yang M, Upshaw B, Storch EA. Development and pilot testing of internet-delivered, family-based cognitive behavioral therapy for anxiety and obsessive-compulsive disorders in autistic youth. J Obsessive Compuls Relat Disord. 2023 Apr;37:100789. doi: 10.1016/j.jocrd.2023.100789. Epub 2023 Feb 14. PMID 36908861